CLINICAL TRIAL: NCT05568706
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of EDP-938 in Non-hospitalized Adults With Acute Respiratory Syncytial Virus Infection Who Are at High Risk for Complications
Brief Title: A Study of EDP-938 in Non-hospitalized Adults With RSV Who Are at High Risk for Complications.
Acronym: RSVHR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDP 938-104
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: RSV Infection
Keywords: High Risk, Respiratory Syncytial Virus
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — EDP-938

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- EDP-938 (Experimental): EDP-938 800 mg, once daily
  Interventions: Drug: EDP-938
- Placebo (Placebo Comparator): Matching placebo, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-938 — Subjects will take EDP-938 once daily for 5 days
  Arms: EDP-938
Drug: Placebo — Subjects will take matching placebo, once daily for 5 days
  Arms: Placebo

SUMMARY:
This is a Phase 2b, randomized, double-blind, placebo-controlled study of EDP-938 administered orally for the treatment of non-hospitalized adult subjects with confirmed RSV infection who are at high risk for complications after RSV infection.

ELIGIBILITY:
Inclusion Criteria:

* At least one of the following conditions that predispose them to complications after RSV infection:

  1. Age ≥65 years
  2. Congestive heart failure (CHF)
  3. Asthma
  4. Chronic obstructive pulmonary disease (COPD)
* The subject has a new onset of any of the following symptom(s) or worsening of pre-existing symptom(s) consistent with a respiratory tract infection no more than 72 hours prior to the administration of the first dose of study drug: feeling feverish, headache, neck pain, fatigue, loss of appetite, interrupted sleep, body aches, sore throat, nasal congestion, cough, cough with phlegm, wheezing, or short of breath.
* The subject reports at least 2 of the following symptoms, one of which must be reported as at least 'moderate' severity: cough, cough with phlegm, wheezing, or short of breath
* The subject has tested positive for RSV infection using a NAAT (polymerase chain reaction [PCR] or other) on a nasal/nasopharyngeal swab sample.
* A woman of childbearing potential who is sexually active with a male must agree to use two effective methods of contraception from the date of Screening until 30 days after her last dose of study drug.
* A male subject who has not had a vasectomy and is sexually active with a woman of childbearing potential must agree to use effective contraception from the date of Screening to 90 days after his last dose of study drug.

Exclusion Criteria:

* The subject has an anticipated need for hospitalization within 24 hours of signing the Study ICF
* The subject receives systemic antiviral, antibacterial, antifungal, or antimycobacterial therapy within 7 days prior to signing the Study ICF
* The subject has concomitant respiratory infections that are viral (other than RSV but including influenza), bacterial, or fungal, including systemic bacterial or fungal infections, within 7 days prior to signing the Study ICF
* The subject has a SARS-CoV-2 test result that is positive within 28 days prior to signing the Study ICF
* The subject has COPD with spirometry results (obtained within 1 year prior to signing the Study ICF) FEV1 ≤35%
* The subject has a known positive human immunodeficiency virus infection, active hepatitis A virus infection, chronic hepatitis B virus infection, and/or current hepatitis C virus (HCV) infection; subjects with a history of HCV infection who have achieved a documented sustained virologic response 12 weeks after completion of HCV therapy may be enrolled.
* The subject has any of the following cardiac conditions: any congenital heart disease, congenital long QT syndrome, or any clinical manifestation resulting in QT interval prolongation
* The subject has immunocompromised status
* The subject is living in institutional care or assisted living facility and is also receiving acute care management for any respiratory condition; Note: Independent living apartments are not considered institutional care or assisted living facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Time to resolution of RSV Lower Respiratory Tract Disease (LRTD) symptoms | Day 1 through Day 33

SECONDARY OUTCOMES:
Time to resolution of LRTD symptoms and 2 systemic symptoms | Day 1 through Day 33
Time to resolution of all RSV symptoms | Day 1 through Day 33
Change from Baseline in severity of RSV LRTD symptoms | Day 1 through Day 33
Change from Baseline for impact scale | Day 1 through Day 33
Time to resolution of Upper Respiratory Tract Disease congestion), LRTD, and 2 systemic symptoms | Day 1 through Day 33
Time to no or mild impact of RSV disease on daily activities, emotions, and social relationships | Day 1 through Day 33
Percentage of participants with post-baseline RSV-related complications | Day 1 through Day 33
Time to improvement in RSV disease | Day 1 through Day 33
Change from Baseline for Health-Related Quality of Life | Day 1 through Day 33
Time to return to usual health | Day 1 through Day 33
Time to return to usual activities | Day 1 through Day 33
Percentage of subjects requiring hospitalization for RSV or other causes; | Day 1 through Day 33
Duration of hospitalization for RSV or other causes | Day 1 through Day 33
All-cause mortality | Day 1 through Day 33
RSV RNA viral load change from Baseline | Days 3, 5, 9, and 14
Change in infectious RSV viral load over time | Up to Day 14
Plasma PK Concentrations of EDP-938 | Up to Day 5
Safety as measured by frequency of adverse events (AEs) | Up to Day 33

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (84):
- United States (31):
  - Voyage Medical, Tempe, Arizona
  - UCSF Fresno, Fresno, California
  - Torrance Clinical Research Institute, Lomita, California
  - Downtown LA Research Center Inc - ClinEdge - PPDS, Los Angeles, California
  - Allianz Research Institute Inc, Westminster, California
  - Allianz Research Institute - Colorado, Aurora, Colorado
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - C&A Clinical Trials Corp, Cape Coral, Florida
  - Beautiful Minds Clinical Research Center, Cutler Bay, Florida
  - Dinamo Research & Diagnostic center, LLC, Hialeah, Florida
  - I.H.S Health LLC, Kissimmee, Florida
  - Dynamic Medical Research, LLC, Miami, Florida
  - Floridian Research Institute, Miami, Florida
  - Orlando VA Healthcare System, Orlando, Florida
  - Ormond Beach Clinical Research, Ormond Beach, Florida
  - CDC Research Institute, LLC, Port Saint Lucie, Florida
  - Research Bay, Inc., Tampa, Florida
  - Santos Research Center, Tampa, Florida
  - Covenant Pulmonary Criticial Care and Research Ins, East Point, Georgia
  - Snake River Research, Idaho Falls, Idaho
  - University of Louisville, Louisville, Kentucky
  - Mercury Street Medical, Butte, Montana
  - Global Health Institute, Syracuse, New York
  - Progressive Medicine of the Triad, LLC, Winston-Salem, North Carolina
  - Toledo Institute of Clinical Research, Toledo, Ohio
  - IMA Clinical Research - Austin - PPDS, Austin, Texas
  - Valley Institute of Research, Fort Worth, Texas
  - HDH Research, Inc., Houston, Texas
  - Metroplex Pulmonary and Sleep Medicine Center-4833 Medical Center Dr Unit 6B, McKinney, Texas
  - SMS Clinical Research, LLC, Mesquite, Texas
  - Eastside Research Associates, Redmond, Washington
- Argentina (7):
  - Instituto Medico Platense, La Plata, Buenos Aires
  - Centro de Investigaciones Medica Mar del Plata, Mar del Plata, Buenos Aires
  - Clinica Privada Independencia, Munro, Buenos Aires
  - Consultorios Médicos Dr. Doreski, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
  - Instituto Del Buen Aire, Santa Fe, Santa Fe Province
  - Clinica Mayo de U.M.C.B. S.R.L, San Miguel de Tucumán, Tucumán Province
- Bulgaria (18):
  - Multiprofile Hospital for Active Treatment Puls AD - PPDS, Blagoevgrad, Blagoevgrad
  - Medical Center For Life EOOD, Burgas, Burgas
  - Diagnostic Consultative Center-1-Sevlievo EOOD, Sevlievo, Gabrovo
  - Medical Center Zdrave-1 OOD, Kozloduy, Kozloduy
  - Medical Center Hera - Kyustendil EOOD, Kyustendil, Kyustendil
  - Specialized Hospital for Active Treatment of Pulmonary Diseases, Troyan Municipality, Lovech
  - Diagnostic Consultative Center 1- Lom EOOD, Lom, Montana
  - Medical Center Hera EOOD, Montana, Montana, Montana
  - Specialized Hospital for Active Treatment of Pulmonary Diseases- Pernik EOOD, Pernik, Pernik
  - Medical Center Prolet EOOD, Rousse, Ruse
  - Medical Center Hipocrena, Sevlievo, Sevlievo
  - Medical Center Hera EOOD, Sofia, Sofia
  - University Multiprofile Hospital for Active Treatment Sofiamed OOD, Sofia, Sofia
  - Medical Center Sanador M EOOD, Sofia, Sofia-Grad
  - Medical Centre Pratia Clinic EOOD Varna, Varna, Varna
  - Medical Center Tara OOD, Veliko Tarnovo, Veliko Tarnovo
  - Specialized Hospital for Active Treatment of Pneumophthisiatric Diseases - Haskovo EOOD, Haskovo
  - Medical Center Neuromedix EOOD, Veliko Tarnovo
- Colombia (6):
  - Servicios de Salud IPS Suramericana S.A.S. - IPS Sura Industriales Medellin, Medellín, Antioquia
  - Clinica de la Costa Ltda - PPDS, Barranquilla, Atlántico
  - Clínica Universidad De la Sabana, Chía, Cundinamarca
  - Fundacion Centro de Investigaciones Clinicas IPS Cardiomet Pereira, Pereira, Risaralda Department
  - Oinsamed S.A.S - Clinica Misericordia, Barranquilla
  - Fundacion Centro de Investigacion Clinica CIC, Medellín
- Czechia (2):
  - MUDr. Jakub Strincl, s.r.o., Liberec, Liberecký kraj
  - Res Medica s.r.o., Nový Knín
- Hospital Miri, Miri, Sarawak, Malaysia
- Mexico (10):
  - Instituto Jalisciense de Investigacion Clinica SA de CV, Guadalajara, Jalisco
  - CICUM San Miguel, Guadalajara, Jalisco
  - Centro de Investigación Clinica Médica y Farmacoló, Guadalajara, Jalisco
  - Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Centro de Atención e Investigación Médica S.A. - México - CAIMED - PPDS, Mexico City, Mexico City
  - Accelerium, S. de R.L. de C.V. - PPDS, Monterrey, Nuevo León
  - Camacho Ortiz, Adrian, Monterrey, Nuevo León
  - Centro de Alta Especialidad Dr. Rafael Lucio, Veracruz, Veracruz
  - FAICIC, Veracruz, Veracruz
  - Oaxaca Site Management Organization - Clinic - OSMO - PPDS, Oaxaca City
- Centrum Medyczne PROFAMILIA, Lodz, Łódź Voivodeship, Poland
- Plucna ambulancia Hrebenar, s.r.o., Spišská Nová Ves, Slovakia
- South Africa (2):
  - Newtown Clinical Research Centre, Johannesburg
  - Be Part Yoluntu Centre, Paarl
- Spain (3):
  - Hospital General Universitario Dr. Balmis, Alicante, Alicante
  - Centro de salud Cabra Matrona Antonia Mesa Fernández, Cabra, Cordoba
  - CHUS - H. Clinico U. de Santiago, Santiago de Compostela
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No